CLINICAL TRIAL: NCT03626792
Title: Effect of Mat Pilates Training on Climacteric Symptoms and Physiological Changes in Women After Menopause
Brief Title: Effect of Mat Pilates Training on Women After Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Jaqueline Pontes Batista, Principal Investigator, Federal University of Uberlandia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68408116.9.0000.5152
Record Dates: First submitted 2017-04-24; First posted 2018-08-13 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Physical Activity; Blood Pressure
Keywords: Pilates; Blood Pressure; Postmenopausal women
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: * Group 1 - Hypertensive: Composed of hypertensive women who participated in a training program with Pilates exercises in the soil associated to the daily antihypertensive of each one.
  * Group 2 - Normotensives: Composed of normotensive women who participated in a training program with solo Pilates exercises without antihypertensive presence.
  Both groups underwent 12 weeks of Pilates training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertensive group (Other): The Mat Pilates session was held lasting 50 minutes of exercises with the first 5 minutes heating and in each exercise performing 10 repetitions with 45 seconds of rest between one exercise and another. For practice, are used only mats, and alternative devices such as the Swiss ball and the flexible ring, as well as body weight and the force of gravity as resistance factors and Borg's subjective perception of effort scale for intensity parameters. The 20 exercises were chosen through the classic exercises thus classified by the creator of the Joseph Pilates method.During the sessions, volunteers were instructed on correct breathing without performing the valsalva maneuver.
  Interventions: Other: Hypertensive group
- Normotensive group (Other): The Mat Pilates session was held lasting 50 minutes of exercises with the first 5 minutes heating and in each exercise performing 10 repetitions with 45 seconds of rest between one exercise and another. For practice, are used only mats, and alternative devices such as the Swiss ball and the flexible ring, as well as body weight and the force of gravity as resistance factors and Borg's subjective perception of effort scale for intensity parameters. The 20 exercises were chosen through the classic exercises thus classified by the creator of the Joseph Pilates method.During the sessions, volunteers were instructed on correct breathing without performing the valsalva maneuver.
  Interventions: Other: Normotensive group

INTERVENTIONS:
Other: Hypertensive group — Pilates 12-week training on the ground, often 3 times a week for 50 minutes of prescribed method exercises.
  Arms: Hypertensive group
Other: Normotensive group — Pilates 12-week training on the ground, often 3 times a week for 50 minutes of prescribed method exercises.
  Arms: Normotensive group

SUMMARY:
This project aims to verify the chronic effect of Mat Pilates exercise on climacteric symptoms, ambulatory blood pressure responses, lipid and glucose profile and pro and anti-inflammatory and antioxidant markers in postmenopausal normotensive and hypertensive women. All volunteers received the same intervention.

DETAILED DESCRIPTION:
The Pilates program was performed three times a week for 12 weeks. Initially a familiarization was made regarding the principles of the method. All volunteers underwent 24-hour blood pressure assessment using ambulatory blood pressure measurement (ABPM) and venous blood samples were collected from fasting, saliva and questionnaires before and after the Pilates training period.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 40 and 70;
* Be post menopausal (amenorrhea for at least 12 months);
* Medical release to perform physical activities.
* Do not present physical problems or cardiovascular complications that prevent the performance of physical exercises;

Exclusion Criteria:

* To present a history of stroke or acute myocardial infarction;
* Smoking;
* Diagnosis of Diabetes Mellitus.
* Present renal pathologies.
* Use medications that interfere with lipid metabolism;
* Use of antihypertensive drugs (except for the hypertensive group);
* Use hormone replacement therapies;
* Present gastrointestinal conditions.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Change from Baseline at 12 weeks
  Resting diastolic and systolic blood pressures will be monitored by Microlife® BP 3BT0A automatic monitor in mmHg.

SECONDARY OUTCOMES:
Ambulatory blood pressure monitoring | Change from Baseline at 12 weeks
  Ambulatory blood pressure monitoring will be monitored during 24 hours using a Dyna+ ABPM device in mmHg.
Kupperman - Blatt Index | Change from Baseline at 12 weeks
  The climacteric symptoms will be evaluated by the following questionnaire Kupperman - Blatt Index. The questionnaire has scores that from 0 to 19 indicate mild symptoms, 20 to 35 moderate and greater than 35 symptoms of severe climacteric.
Cervical Scale | Change from Baseline at 12 weeks
  The climacteric symptoms will be evaluated by the following questionnaire Cervical Scale. The questionnaire does not have scales. Indicates only a high or low score regarding the presence of climacteric symptoms.
Menopause Rating Scale (MRS) | Change from Baseline at 12 weeks
  The climacteric symptoms will be evaluated by the following questionnaire Menopause Rating Scale (MRS). The scores from 0 to 4 of the questionnaire indicate absence of symptoms, as well as from 5 to 8 presence of mild symptoms, 9 to 15 moderate and greater than 16 symptoms of severe climacteric.
Sleep quality | Change from Baseline at 12 weeks
  Sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI).A score of 0 to 4 indicates a good quality of sleep, 5 to 10 quality of bad sleep and greater than 10 the presence of sleep disorder.

OTHER OUTCOMES:
Biochemical analyzes | Change from Baseline at 12 weeks
  From the serum and/or plasma and saliva samples collected and stored, analyzes for lipid profile (total cholesterol and fractions, and triglycerides) and glycemia at rest and for the concentrations of inflammatory cytokines and changes in the activity of the Antioxidant system.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Puga, Phd, Study Director — Federal University of Uberlandia
Locations (1):
- Jaqueline Pontes Batista, Uberlândia, Minas Gerais, Brazil